CLINICAL TRIAL: NCT01168453
Title: Changes in the Relationship Between the Right Internal Jugular Vein and Anatomical Landmark After Head Rotation
Brief Title: Changes in Anatomical Landmark Locations
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Soonchunhyang University Hospital, President of Soonchunhyang University Hospital
Other Study IDs: LoIJV
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-07

CONDITIONS: Anesthesia, General; Intubation
Keywords: jugular vein; anatomy; ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- neutral head position: supine with neutral head position
  Interventions: Behavioral: head position change
- head rotation: supine with 30° head rotation
  Interventions: Behavioral: head position change

INTERVENTIONS:
Behavioral: head position change — AL-US distance measure using the ultrasound in two different head position

SUMMARY:
This study was performed to ultrasonographically demonstrate the changes in relationship between the right internal jugular vein (IJV) and an anatomical landmark in two different head positions: neutral and rotational.

DETAILED DESCRIPTION:
Background: This study was performed to ultrasonographically demonstrate the changes in relationship between the right IJV and an anatomical landmark in two different head positions: neutral and rotational.

Methods: One hundred patients scheduled for elective surgery under general anesthesia with endotracheal intubation were enrolled in this study. The patients were placed in the supine position with a neutral head position and without a pillow. The apex of the triangle formed by the sternal and clavicular heads of the sternocleidomastoid muscle and clavicle was marked (anatomical landmark point: AL point). The ultrasonography of the neck anatomy was performed, and a mark was placed at the central point of the IJV to the skin (ultrasonography point: US point). The other investigator measured the distances from the AL point to the US point (AL-US distance). The patient's head was then turned 30° to the left; the same procedure was repeated and the AL-US distance was again measured. The changes in AL-US distance were calculated.

ELIGIBILITY:
Inclusion Criteria:

* 100 patients weighing 40 - 100 kg and with heights of 140 - 190 cm

Exclusion Criteria:

* a history of neck surgery or trauma involving the neck, previous IJV-related interventions (e.g., venous catheterization), limitation of neck movement, and a body mass index ≥ 30.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery under general anesthesia with endotracheal intubation, were enrolled in the study between May 2009 and February 2010.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
anatomical landmark point (AL) - ultrasonography point (US) distance(the distances from the AL point to the US point ) | within 5 minutes after itubation
  The distance between the two points was considered "positive" if the US point was lateral to the AL point and "negative" if it was medial to the AL point.

SECONDARY OUTCOMES:
The average depth of the right IJV | within 5 minutes after intubation
  measure the depth of the right IJV center in ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Park, Dr., Study Chair — Soonchuhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea